CLINICAL TRIAL: NCT00099762
Title: Selective Venous Catheterization for the Localization of Phosphaturic Mesenchymal Tumors
Brief Title: Catheterization to Locate Mesenchymal Tumors in Patients With Tumor-Induced Osteomalacia or Oncogenic Osteomalacia
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050050; 05-D-0050
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-02

CONDITIONS: Osteomalacia; Neoplasms
Keywords: Tumor Induced Osteomalacia; FGF-23; Phosphatonin; Hypophosphatemia; Oncogenic Osteomalacia; Phosphaturic Mesenchymal Tumor; TIO; Osteogenic Osteomalacia; OOM
MeSH Terms: conditions — Osteomalacia; Neoplasms; Oncogenic osteomalacia; Hypophosphatemia

SUMMARY:
This study will use a procedure called selective venous catheterization in patients with tumor-induced osteomalacia (TIO) or oncogenic osteomalacia (OOM) to try to locate very small tumors that produce proteins called phosphatonins. Too much phosphatonin in the blood causes the kidneys to allow large amounts of phosphorus to be excreted in the urine, leading to low blood levels of phosphorus and, in turn, to osteomalacia (a condition of soft bones). Osteomalacia can cause bone fractures requiring many surgical procedures that can leave patients in pain. Patients may also feel weak and can lose height from massive bone loss. Selective venous catheterization is a way to measure the amount of phosphatonin in the blood and may be used as a way to locate phosphatonin-producing tumors that cannot be found using standard imaging techniques.

Patients with TIO or OOM are screened under NIDR Protocol 01-D-0184 with a medical history, review of medical records and routine physical examination. Other procedures may include blood tests, urine tests, and imaging tests, such as x-rays, bone densitometry, bone scan, computed tomography (CT) and magnetic resonance imaging (MRI). This study will include mostly patients whose tumors were not able to be located through imaging procedures, but also a few patients whose tumors were located.

All participants, regardless of whether or not their tumor was located, undergo selective venous catheterization. For this procedure, a radiologist inserts a catheter (thin flexible tube) into the body and uses fluoroscopy (a type of x-ray) to guide the tip of the catheter to different places in the body to collect small amounts of blood from the different areas. After the procedure, the patient lies flat for 2 hours and avoids moving his or her leg on the side where the catheter was placed.

The blood is analyzed to measure the amount phosphatonin is in each sample, and the amounts are compared to the average amount of phosphatonin in the general blood circulation. If a higher level of phosphatonin is found in one area and the location of the tumor is unknown, the patient undergoes imaging in that area. If a tumor is found and it is in an area where it can be removed surgically, the patient is given the option to have the surgery. If the tumor is not found by imaging done after the first catheterization procedure, the patient has the option to have a second catheterization, taking samples of blood only from the area where the phosphatonin was found to be the highest during the sampling procedure.

DETAILED DESCRIPTION:
Phosphaturic mesenchymal tumors elaborate phosphate lowering factors (phosphatonins) which lead to tumor induced osteomalacia/osteogenic osteomalacia (TIO/OOM). Patients with TIO/OOM suffer years of significant morbidity and debilitation unless their tumors, which are notoriously difficult to locate, are removed.

Selective venous catheterization has been used to localize hormonally active neoplasms by demonstrating a gradient in the concentration of the hormone of interest between the vessel immediately draining the tumor site and the peripheral circulation. The primary objective of this protocol is to evaluate the utility of combining selective venous catheterization with biochemical assays that identify phosphatonins in the serum as a way to identify phosphatonin gradients and thereby localize phosphaturic tumors.

Our study population will consist of TIO/OOM patients with non-localized phosphaturic tumors as well as five patients whose lesions have been identified with some certainty by conventional imaging techniques. These individuals will undergo selective venous catheterization during which blood samples will be obtained and processed for the presence of phosphatonins. The primary endpoint will be met if a gradient indicating a possible tumor is found, focused clinical imaging in the appropriate anatomical sub-region identifies a lesion, and the lesion is confirmed to be a phosphaturic mesenchymal tumor upon surgical removal.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have the clinical diagnosis of TIO/OOM to be considered for enrollment in this study. The diagnosis will be based upon a clinical history including some or all of: rickets (children), pathological fractures, bone pain, muscle weakness, low serum phosphorus with concomitant inappropriately high urine phosphorus, low or inappropriately low-normal serum vitamin 1,25 (OH)(2)-vitamin D3, and an elevated FGF-23 level in the absence of a family history of a phosphate wasting syndrome. Along with the clinical symptoms listed above, the patient must have undergone routine clinical imaging.

Inclusion will be limited to all patients in whom a likely lesion was not localized by imaging, plus five patients for whom a likely lesion has been identified by imaging. Patients with a likely lesion identified will serve as positive controls.

Patients must be able to give informed consent.

EXCLUSION CRITERIA:

Patients with co-morbidities that would increase the risk of selective venous catheterization will be excluded from the study. This includes but is not limited to medical conditions such as: poorly controlled diabetes, renal insufficiency, chronic obstructive pulmonary disease, anemia, hypertension, clotting disorders, etc.

Pregnancy is a contraindication to this venous catheterization procedure. A serum Beta-Hcg will be required for all eligible women of childbearing age unless documentation of a hysterectomy or other condition that makes pregnancy impossible is provided.

Inability or unwillingness to give informed consent will exclude patients from this study. Female patients who will not allow pregnancy testing and will not provide documentation indicating a medical condition that makes pregnancy impossible will not be eligible for this study.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 2004-12-15; Primary Completion 2009-09-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] ADHR Consortium. Autosomal dominant hypophosphataemic rickets is associated with mutations in FGF23. Nat Genet. 2000 Nov;26(3):345-8. doi: 10.1038/81664. PMID 11062477
- [Background] Berndt T, Craig TA, Bowe AE, Vassiliadis J, Reczek D, Finnegan R, Jan De Beur SM, Schiavi SC, Kumar R. Secreted frizzled-related protein 4 is a potent tumor-derived phosphaturic agent. J Clin Invest. 2003 Sep;112(5):785-94. doi: 10.1172/JCI18563. PMID 12952927
- [Background] Bowe AE, Finnegan R, Jan de Beur SM, Cho J, Levine MA, Kumar R, Schiavi SC. FGF-23 inhibits renal tubular phosphate transport and is a PHEX substrate. Biochem Biophys Res Commun. 2001 Jun 22;284(4):977-81. doi: 10.1006/bbrc.2001.5084. PMID 11409890